CLINICAL TRIAL: NCT02667912
Title: Anatomically Optimized Distal Renal Denervation for Treatment of Resistant Hypertension
Brief Title: Distal Renal Denervation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tomsk National Research Medical Center of the Russian Academy of Sciences (Other)
Responsible Party: Principal Investigator, Stanislav Pekarskiy, Principal Investigator, Tomsk National Research Medical Center of the Russian Academy of Sciences
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 022
Record Dates: First submitted 2016-01-26; First posted 2016-01-29 (Estimated); Results first posted 2019-02-01 (Actual); Last update posted 2021-10-25 (Actual); Status verified 2021-10

CONDITIONS: Hypertension, Resistant to Conventional Therapy
Keywords: Hypertension, Catheter Ablation, Renal Nerves
MeSH Terms: conditions — Hypertension Resistant to Conventional Therapy; Hypertension

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Distal renal denervation (Experimental): Endovascular denervation of segmental branches of renal artery
  Interventions: Procedure: Distal renal denervation
- Conventional renal denervation (Active Comparator): Endovascular denervation of main trunk of renal artery
  Interventions: Procedure: Conventional renal denervation

INTERVENTIONS:
Procedure: Distal renal denervation — Percutaneous endovascular intervention when catheter-based electrode (Symplicity Flex; Medtronic, Inc.) is used for stepwise radiofrequency energy delivery to segmental branches of the renal artery in a number of points distributed along the length and circumference of the vessels in order to ablate renal nerve plexus
  Arms: Distal renal denervation
Procedure: Conventional renal denervation — Percutaneous endovascular intervention when catheter-based electrode (Symplicity Flex; Medtronic, Inc.) is used for stepwise radiofrequency energy delivery to the main trunk of the renal artery in a number of points equally distributed along its length and circumference in order to ablate renal nerve plexus
  Arms: Conventional renal denervation

SUMMARY:
Objective of this study is to evaluate whether a distal mode of endovascular renal denervation with the treatment performed primarily in segmental branches of renal artery is more effective than conventional mode of the intervention with the treatment equally distributed within its main trunk for the treatment of drug-resistant hypertension.

DETAILED DESCRIPTION:
Recent spectacular failure of renal denervation (RDN) therapy in SymplicityHTN-3 trial in fact might be easily predicted from the very beginning. Conventional RDN done as 4-6 point treatments equally distributed within main trunk of renal artery (RA) may only be effective if renal plexus tightly surrounds the artery throughout its whole course with equal longitudinal and circumferential density of the nerve fibers. While this idea itself is unnaturally idealistic also a number of surgical studies demonstrated that proximally majority of renal nerves go at a distance from RA obliquely to its course and join the artery mainly in its distal part (fan-shaped renal plexus with wide base directed toward aorta and apex converging to renal gate). We developed a distal mode of RDN targeting segmental branches of RA and conducted a single-center double-blind randomized controlled parallel group study to compare its efficacy and safety to those of conventional RDN in patients with drug-resistant hypertension.

ELIGIBILITY:
Inclusion Criteria:

* systolic BP is equal or greater than 160 mmHg or diastolic BP is equal or greater than 100 mmHg,
* stable (>3 months) treatment with full doses of at least 3 antihypertensive drugs including a diuretic,
* given written informed consent

Exclusion Criteria:

* secondary hypertension
* 24h-mean systolic BP <135 mmHg,
* estimated glomerular filtration rate (eGFR) < 30 mL/min/1.73 m2,
* extended disease of renal artery,
* any other clinically important disorders/comorbidities significantly increasing risk of endovascular intervention (investigator's assessment)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2013-01; Primary Completion 2016-07 (Actual); Study Completion 2016-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stanislav Pekarskiy, MD, PhD, Principal Investigator — Tomsk National Research Medical Center of the Russian Academy of Sciences
Locations (1):
- Tomsk National Research Medical Center of the Russian Academy of Sciences, Tomsk, Russia

REFERENCES:
- [Result] Pekarskiy SE, Baev AE, Mordovin VF, Semke GV, Ripp TM, Falkovskaya AU, Lichikaki VA, Sitkova ES, Zubanova IV, Popov SV. Denervation of the distal renal arterial branches vs. conventional main renal artery treatment: a randomized controlled trial for treatment of resistant hypertension. J Hypertens. 2017 Feb;35(2):369-375. doi: 10.1097/HJH.0000000000001160. PMID 28005705
- [Derived] Pisano A, Iannone LF, Leo A, Russo E, Coppolino G, Bolignano D. Renal denervation for resistant hypertension. Cochrane Database Syst Rev. 2021 Nov 22;11(11):CD011499. doi: 10.1002/14651858.CD011499.pub3. PMID 34806762

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Distal Renal Denervation | Conventional Renal Denervation
Started | 28 | 27
Six Months | 27 | 24
Completed | 23 | 24
Not Completed | 5 | 3
Not completed — Death | 3 | 1
Not completed — Withdrawal by Subject | 1 | 2
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Distal Renal Denervation | Conventional Renal Denervation | Total
Number analyzed (Participants) | 28 | 27 | 55
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.5 (9.4) | 57.3 (9.5) | 56.9 (9.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 17 | 35
  Male | 10 | 10 | 20
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 2 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 27 | 25 | 52
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Russia | 28 | 27 | 55
Concomitant coronary artery disease (CAD) [Count of Participants; unit: Participants] | 12 | 12 | 24
Concomitant diabetes [Count of Participants; unit: Participants] | 14 | 13 | 27
A number of antihypertensive drugs taken [Mean (Standard Deviation); unit: Medication (single active ingredient)] | 4.1 (1.1) | 4.3 (0.9) | 4.2 (1.0)
A use of diuretics [Count of Participants; unit: Participants] | 27 | 27 | 54
Office systolic BP [Mean (Standard Deviation); unit: mmHg] | 170.8 (23.0) | 169.4 (23.6) | 170.1 (23.1)
Office diastolic BP [Mean (Standard Deviation); unit: mmHg] | 93.4 (17.3) | 94.2 (19.6) | 93.8 (18.3)
24-hour systolic BP [Mean (Standard Deviation); unit: mmHg] | 168.0 (24.1) | 158.0 (15.2) | 162.6 (20.6)
24-hour diastolic BP [Mean (Standard Deviation); unit: mmHg] | 91.6 (19.1) | 88.0 (19.6) | 89.6 (18.2)
Left ventricular mass [Mean (Standard Deviation); unit: g] | 260.3 (68.6) | 259.8 (84.5) | 260.1 (76.1)
24-hour proteinuria [Mean (Standard Deviation); unit: g] | 0.12 (0.19) | 0.16 (0.30) | 0.15 (0.25)
Serum creatinine [Mean (Standard Deviation); unit: mMol/L] | 79.3 (24.0) | 89.4 (20.7) | 84.2 (22.8)
estimated glomerular filtration rate (eGFR) [Mean (Standard Deviation); unit: ml/min/m2] — Glomerular filtration rate estimated using Modification of Diet in Renal Disease (MDRD) Study formula
  ml/min/m2 | 79.3 (24.0) | 70.6 (13.1) | 77.3 (20.0)

OUTCOME MEASURES:

1. Primary Outcome: Changes of 24h-mean Systolic BP Assessed by Ambulatory Blood Pressure Monitoring (ABPM)
Time Frame: From baseline to 6 months
Population: The subjects who completed 6 months follow up without serious violations of the study protocol - per protocol set
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Distal Renal Denervation | Conventional Renal Denervation
Number analyzed (Participants) | 27 | 24
mmHg | 21.1 (19.3) | 10.3 (17.8)
Statistical Analysis 1: Comparison: Distal Renal Denervation vs Conventional Renal Denervation; Test type: Superiority; p = 0.045, t-test, 2 sided — The a priori threshold for statistical significance <0.05; Mean Difference (Final Values) = 10.8, 95% CI 2-sided [0.3 to 21.4]

2. Secondary Outcome: Number of Adverse Events
Time Frame: From baseline to 6 months
Measure: Number; unit: adverse event
Arm/Group | Distal Renal Denervation | Conventional Renal Denervation
Number analyzed (Participants) | 27 | 24
adverse event | 1 | 0

3. Secondary Outcome: Number of Adverse Events
Time Frame: From baseline to 12 months
Population: A baseline population except those who refused to continue in the study before final assessment and thereby whose status was unknown at 12 months follow up (5 in the distal denervation arm and 3 patients in conventional denervation arm).
Measure: Number; unit: adverse event
Arm/Group | Distal Renal Denervation | Conventional Renal Denervation
Number analyzed (Participants) | 23 | 24
adverse event | 4 | 2

4. Secondary Outcome: Changes of Arterial Resistance Index Measured by Doppler Flowmetry in the Right Segmental Renal Arteries
Description: Resistance index is calculated as the relative difference between a peak systolic and end diastolic blood flow velocities assessed by ultrasound Doppler flowmetry
Time Frame: From baseline to 6 months
Population: Per protocol set (PPS)
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Distal Renal Denervation | Conventional Renal Denervation
Number analyzed (Participants) | 25 | 19
ratio | 0.018 (0.064) | 0.017 (0.058)
Statistical Analysis 1: Comparison: Distal Renal Denervation vs Conventional Renal Denervation; Test type: Superiority; p = 0.96, t-test, 2 sided

5. Secondary Outcome: Changes of Arterial Resistance Index Measured by Doppler Flowmetry in the Left Segmental Renal Arteries
Description: Resistance index calculated as the relative difference between a peak systolic and end diastolic blood flow velocities assessed by ultrasound Doppler flowmetry
Time Frame: From baseline to 6 months
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Distal Renal Denervation | Conventional Renal Denervation
Number analyzed (Participants) | 25 | 19
ratio | 0.006 (0.066) | 0.032 (0.066)
Statistical Analysis 1: Comparison: Distal Renal Denervation vs Conventional Renal Denervation; Test type: Other; p = 0.203, t-test, 2 sided

6. Secondary Outcome: Changes of Serum Creatinine
Time Frame: From baseline to 6 months
Measure: Mean (Standard Deviation); unit: μmol/l
Arm/Group | Distal Renal Denervation | Conventional Renal Denervation
Number analyzed (Participants) | 23 | 23
μmol/l | 2.0 (13.4) | 2.3 (12.5)
Statistical Analysis 1: Comparison: Distal Renal Denervation vs Conventional Renal Denervation; Test type: Superiority; p = 0.27, t-test, 2 sided; Mean Difference (Final Values) = -4.3, 95% CI 2-sided [-11.9 to 3.4]

7. Secondary Outcome: Changes of Serum Creatinine
Time Frame: From baseline to 12 months
Population: Intention-to-treat (ITT) analysis by Last Observation Carried Forward (LOCF) method. (Six month data were used in 4 late (>6 months) dropouts and also in 1 patient without 12 month' ABPM, 1 month data were used in 2 early (<6 months) dropouts. One patient had no post procedure data at all and was excluded from analysis)
Measure: Mean (Standard Error); unit: μmol/l
Arm/Group | Distal Renal Denervation | Conventional Renal Denervation
Number analyzed (Participants) | 24 | 24
μmol/l | 9.8 (19.7) | 2.0 (19.8)
Statistical Analysis 1: Comparison: Distal Renal Denervation vs Conventional Renal Denervation; Test type: Superiority; p = 0.17, t-test, 2 sided — The a priori threshold for statistical significance p<0.05; Mean Difference (Final Values) = 7.8, 95% CI 2-sided [-3.7 to 19.3], Standard Error of Mean 5.7

8. Secondary Outcome: Changes of Estimated Glomerular Filtration Rate (eGFR)
Time Frame: From baseline to 6 months
Population: The subjects with available data
Measure: Mean (Standard Deviation); unit: ml/min/square meter
Arm/Group | Distal Renal Denervation | Conventional Renal Denervation
Number analyzed (Participants) | 28 | 26
ml/min/square meter | 7.6 (13.6) | 1.3 (12.5)

9. Secondary Outcome: Changes of Estimated Glomerular Filtration Rate (eGFR)
Time Frame: From baseline to 12 months
Population: ITT analysis by Last Observation Carried Forward (LOCF) method in the subjects with the available data. (Six month data were used in 4 late (>6 months) dropouts and also in 1 patient without 12 month' ABPM, 1 month data were used in 2 early (<6 months) dropouts. One patient had no post procedure data at all and was excluded from analysis)
Measure: Mean (Standard Deviation); unit: ml/min/square meter
Arm/Group | Distal Renal Denervation | Conventional Renal Denervation
Number analyzed (Participants) | 25 | 24
ml/min/square meter | -7.6 (13.6) | -1.3 (12.5)

10. Secondary Outcome: Changes of 24h-mean Diastolic BP
Time Frame: From baseline to 6 months
Population: PPS
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Distal Renal Denervation | Conventional Renal Denervation
Number analyzed (Participants) | 27 | 24
mmHg | 11.1 (11.9) | 7.0 (10.6)
Statistical Analysis 1: Comparison: Distal Renal Denervation vs Conventional Renal Denervation; Test type: Superiority; p = 0.213, t-test, 2 sided

11. Secondary Outcome: Changes of 24h-mean Systolic BP
Time Frame: From baseline to 12 months
Population: ITT analysis by Last Observation Carried Forward (LOCF) method in the subjects with the available data . (Six month data were used in 4 late (>6 months) dropouts and also in 1 patient without 12 month' ABPM, 1 month data were used in 2 early (<6 months) dropouts. One patient had no post procedure data at all and was excluded from analysis)
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Distal Renal Denervation | Conventional Renal Denervation
Number analyzed (Participants) | 28 | 26
mmHg | 22.1 (20.6) | 11.5 (16.4)
Statistical Analysis 1: Comparison: Distal Renal Denervation vs Conventional Renal Denervation; Test type: Superiority; p = 0.041, t-test, 2 sided

12. Secondary Outcome: Changes of 24h-mean Diastolic BP
Time Frame: From baseline to 12 months
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Distal Renal Denervation | Conventional Renal Denervation
Number analyzed (Participants) | 28 | 26
mmHg | 11.2 (12.3) | 7.9 (10.6)
Statistical Analysis 1: Comparison: Distal Renal Denervation vs Conventional Renal Denervation; Test type: Other; p = 0.304, t-test, 2 sided

13. Secondary Outcome: Changes of Office Systolic BP
Time Frame: From baseline to 6 months
Population: PPS
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Distal Renal Denervation | Conventional Renal Denervation
Number analyzed (Participants) | 27 | 24
mmHg | 26.1 (226.8) | 21.2 (23.3)
Statistical Analysis 1: Comparison: Distal Renal Denervation vs Conventional Renal Denervation; Test type: Superiority; p = 0.49, t-test, 2 sided

14. Secondary Outcome: Changes of Office Systolic BP
Time Frame: From baseline to 12 months
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Distal Renal Denervation | Conventional Renal Denervation
Number analyzed (Participants) | 28 | 26
mmHg | 12.8 (15.7) | 10.8 (18.8)
Statistical Analysis 1: Comparison: Distal Renal Denervation vs Conventional Renal Denervation; Test type: Superiority; p = 0.66, t-test, 2 sided

15. Secondary Outcome: Changes of Office Diastolic BP
Time Frame: From baseline to 6 months
Population: PPS
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Distal Renal Denervation | Conventional Renal Denervation
Number analyzed (Participants) | 27 | 24
mmHg | 12.6 (15.6) | 10.4 (12.1)
Statistical Analysis 1: Comparison: Distal Renal Denervation vs Conventional Renal Denervation; Test type: Superiority; p = 0.59, t-test, 2 sided

16. Secondary Outcome: Changes of Office Diastolic BP
Time Frame: From baseline to 12 months
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Distal Renal Denervation | Conventional Renal Denervation
Number analyzed (Participants) | 28 | 26
mmHg | 12.8 (15.7) | 10.8 (18.8)
Statistical Analysis 1: Comparison: Distal Renal Denervation vs Conventional Renal Denervation; Test type: Superiority; p = 0.66, t-test, 2 sided

17. Secondary Outcome: Changes of Daytime Systolic BP
Time Frame: From baseline to 6 months
Population: PPS
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Distal Renal Denervation | Conventional Renal Denervation
Number analyzed (Participants) | 26 | 24
mmHg | 22.2 (19.9) | 10.9 (18.9)
Statistical Analysis 1: Comparison: Distal Renal Denervation vs Conventional Renal Denervation; Test type: Superiority; p = 0.04, t-test, 2 sided

18. Secondary Outcome: Changes of Daytime Mean Systolic BP
Time Frame: From baseline to 12 months
Population: ITT analysis by Last Observation Carried Forward (LOCF) method. (Six month data were used in 4 late (>6 months) dropouts and also in 1 patient without 12 month' ABPM, 1 month data were used in 2 early (<6 months) dropouts. One patient had no post procedure data at all and was excluded from analysis)
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Distal Renal Denervation | Conventional Renal Denervation
Number analyzed (Participants) | 28 | 26
mmHg | 22.1 (20.5) | 11.5 (18.6)
Statistical Analysis 1: Comparison: Distal Renal Denervation vs Conventional Renal Denervation; Test type: Superiority; p = 0.054, t-test, 2 sided

19. Secondary Outcome: Changes of Daytime Mean Diastolic BP
Time Frame: From baseline to 6 months
Population: PPS
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Distal Renal Denervation | Conventional Renal Denervation
Number analyzed (Participants) | 26 | 24
mmHg | 11.8 (12.9) | 10.9 (18.9)
Statistical Analysis 1: Comparison: Distal Renal Denervation vs Conventional Renal Denervation; Test type: Superiority; p = 0.204, t-test, 2 sided

20. Secondary Outcome: Changes of Daytime Mean Diastolic BP
Time Frame: From baseline to 12 months
Population: ITT analysis by Last Observation Carried Forward (LOCF). (Six month data were used in 4 late (>6 months) dropouts and also in 1 patient without 12 month' ABPM, 1 month data were used in 2 early (<6 months) dropouts. One patient had no post procedure data at all and was excluded from analysis)
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Distal Renal Denervation | Conventional Renal Denervation
Number analyzed (Participants) | 28 | 26
mmHg | 11.3 (12.6) | 7.9 (12.3)
Statistical Analysis 1: Comparison: Distal Renal Denervation vs Conventional Renal Denervation; Test type: Superiority; p = 0.324, t-test, 2 sided

21. Secondary Outcome: Changes of Nighttime Mean Systolic BP
Time Frame: From baseline to 6 months
Population: PPS
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Distal Renal Denervation | Conventional Renal Denervation
Number analyzed (Participants) | 26 | 24
mmHg | 16.5 (19.7) | 9.3 (20.9)
Statistical Analysis 1: Comparison: Distal Renal Denervation vs Conventional Renal Denervation; Test type: Superiority; p = 0.217, t-test, 2 sided

22. Secondary Outcome: Changes of Nighttime Mean Systolic BP
Time Frame: From baseline to 12 months
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Distal Renal Denervation | Conventional Renal Denervation
Number analyzed (Participants) | 27 | 26
mmHg | 17.8 (22.0) | 10.9 (19.2)
Statistical Analysis 1: Comparison: Distal Renal Denervation vs Conventional Renal Denervation; Test type: Superiority; p = 0.238, t-test, 2 sided

23. Secondary Outcome: Changes of Nighttime Mean Diastolic BP
Time Frame: From baseline to 6 months
Population: PPS
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Distal Renal Denervation | Conventional Renal Denervation
Number analyzed (Participants) | 26 | 24
mmHg | 6.7 (12.8) | 6.5 (11.8)
Statistical Analysis 1: Comparison: Distal Renal Denervation vs Conventional Renal Denervation; Test type: Superiority; p = 0.969, t-test, 2 sided

24. Secondary Outcome: Changes of Nighttime Mean Diastolic BP
Time Frame: From baseline to 12 months
Population: ITT analysis by Last Observation Carried Forward (LOCF) method in the subjects with the available data. (6 month data were used in 4 late (>6 months) dropouts and also in 1 patient without 12 month' ABPM, 1 month data were used in 2 early (<6 months) dropouts. One patient had no post procedure data at all and was excluded from analysis)
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Distal Renal Denervation | Conventional Renal Denervation
Number analyzed (Participants) | 27 | 26
mmHg | 7.2 (12.5) | 7.5 (12.1)
Statistical Analysis 1: Comparison: Distal Renal Denervation vs Conventional Renal Denervation; Test type: Superiority; p = 0.37, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: 6 months
Description: Serious Adverse Events
Arm/Group | Distal Renal Denervation | Conventional Renal Denervation
Serious Adverse Events (participants affected / at risk) | 1/27 | 0/24
Other Adverse Events (participants affected / at risk) | 0/27 | 0/24
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Distal Renal Denervation (N=27) | Conventional Renal Denervation (N=24)
Post-punctional pseudoaneuryzm (Surgical and medical procedures) | 1 (1) | 0 (0) — Hemorrhage from the femoral artery at the punction site after removal of intra-arterial introducer

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes